CLINICAL TRIAL: NCT01510197
Title: Identification of a Risk Profile in Patients With Atrial Fibrillation
Brief Title: Risk Profile for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, I.C. Van Gelder, MD, PhD, University Medical Center Groningen
Other Study IDs: Biomarker
Record Dates: First submitted 2012-01-01; First posted 2012-01-16 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Arrhythmia; Rhythm control
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to assess the risk profile in patients with atrial fibrillation, which represents the degree of changes (remodeling) in the atrial tissue and which can help to predict in which patients rhythm control will be successful. This risk profile will consist of a combination of underlying (heart) disease and risk factors, as measured with use of parameters obtained with echocardiography, circulating biomarkers and other relevant clinical data. Ultimately this risk profile can be used to guide type of (rhythm) control therapy in individual patients with atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation is responsible for substantial morbidity and mortality.Identification of patients with AF that is difficult to treat may improve the outcome of rhythm control therapy. Left atrial size or volume could be a useful tool to select patients that will benefit from rhythm control therapy.Beside echocardiographic parameters,atrial fibrillation has been also associated with circulating biomarkers in blood like collagen metabolism, inflammatory mediators,neurohumoral factors and proteins/proteomic profiles. Beside more accepted risk factors (myocardial ischemia, diabetes and pulmonary disease)other less well-known clinical factors (sleep apnea, alcohol or other intoxication abuse, excessive physical activity, esophageal problems and increased body mass index) may also predict the outcome of rhythm control.It seems also plausible that recurrent atrial fibrillation within one month after start of rhythm control is associated with a different risk profile than late atrial fibrillation recurrences.During this study we will try to identify patients with atrial fibrillation who are more or less likely to respond to rhythm control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Short-lasting symptomatic paroxysmal or persistent AF;
* Rhythm control strategy is preferred;
* No contra-indication for oral anticoagulation;
* Age > 18 years;
* Written informed consent

Exclusion Criteria:

* Total history of heart failure and/ or of severe valvular disease > 3 years;
* Severe valvular disease;
* Acute coronary syndrome/ myocardial infarction/ percutaneous coronary intervention/ coronary artery bypass surgery within the past one month;
* Post-operative AF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with short-lasting symptomatic paroxysmal or persistent AF
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
assess the risk profile associated with success of rhythm control therapy at follow-up. | 12 months
  1) < 1 second AF on end-of-study ECG; (2) < 30 seconds AF on end-of-study 48-hour Holter recording

SECONDARY OUTCOMES:
Time to recurrence of (a)symptomatic AF; | 1+12+60 months
  by assessment Percentage AF-burden on 24-Holter during follow up
Failure of rhythm control, i.e. permanent AF; | 1+12+60 months
  <1 second AF on ECG during rhythm control medication or after electric cardioversion.
Risk profiles associated with early versus late AF recurrence; | 1+12+60 months
  Parameters including underlying (heart) disease and risk factors (age, family history for AF, signs of ischemia, coronary risk factors, pulmonary disease, diabetes, obesity, sleep apnea, esophageal problems), lifestyle (caffeine and alcohol intake, exercise), autonomic trigger patterns of AF (i.e. vagal or adrenergic induced AF, or combination)
Progression of paroxysmal AF to persistent or permanent AF and of persistent AF to permanent AF | 1+12+60 months
  3-lead Holter monitoring will be used
Changes in atrial and ventricular echocardiographic parameters | 1+12+60 month
  Echocardiographic measures of LA size (LA size parasternal long axis view, LA volume,LA ejection fraction measurement, electro-echocardiographic parameters (Tissue Doppler total atrial conduction time (during sinus rhythm), AF cycle length and velocity (during AF)), and parameters of diastolic dysfunction, including E (early mitral valve flow velocity), A (late mitral valve flow velocity), E/A ratio, deceleration time, E' (early tissue Doppler lengthening velocity), and E/E' ratio
Cardiovascular morbidity and mortality | 1+12+60 months
  hospitalization for cardiovascular reasons, non-cardiovascular and cardiovascular death will be carefully monitored through-out the study.
Pulmonary vein ablation | 1+12+60 months
  hospital admission for pulmonary vein ablation will be monitoring during the study.
Differences in clinical profile and outcome between patients presenting at the emergency room and the outpatient department | Baseline,12+60 months
  collected parameters will be compared between these two groups.
relate risk profiles to quality of life | 1+12+60 months
  a quality of life questionnaire will be handed
biomarkers associated with success of rhythm control | baseline, 12 months, 60 months
  biomarker profiles (collagen mediated, inflammation, neurohumoral) associated with underlying mechanism of AF

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C van Gelder, Md PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical center Groningen, Groningen, Provincie Groningen, Netherlands